CLINICAL TRIAL: NCT05059054
Title: Effectiveness of Strengthening Exercise Program Compare With Foot Orthoses in Patients With Plantar Heel Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mahidol University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2020/285.2109
Record Dates: First submitted 2021-06-21; First posted 2021-09-28 (Actual); Last update posted 2023-03-15 (Actual); Status verified 2023-03

CONDITIONS: Plantar Fascitis; Fasciitis, Plantar, Chronic
Keywords: Plantar Fasciitis; Strength Training; Foot Orthosis
MeSH Terms: conditions — Fasciitis, Plantar | interventions — Population Groups

STUDY DESIGN:
Intervention Model Description: Comparison between the exercise program and insole program.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Strengthening group (Experimental): Strengthening exercise
  Interventions: Other: Strengthening exercise
- Insole group (Active Comparator): Insole application
  Interventions: Other: Insole (CFO) group

INTERVENTIONS:
Other: Strengthening exercise — Strengthening exercise program Participants performed this protocol at home for 3 times per day. The participants progress their exercise based on the achievement of the previous level of each exercise protocol. The physical therapist recorded the level of each exercise for each participant during eight times of treatment. Total time for this section is approximately 30 minutes. Detail of the strengthening exercise is in the following.
  1. Toe curl exercise (toe flexors strengthening)
  2. Ankle evertor exercise (peroneal strengthening)
  3. Ankle invertor exercise (tibialis posterior strengthening)
  4. Heel raise exercise (high-load strength training)
  Arms: Strengthening group
Other: Insole (CFO) group — The CFO insole group The participants will receive the foot assessment before making the CFO for each participant. The 3-quarter-length CFO will be made from thermoplastic material (rigid foot orthoses) which consists of four layers i.e. two layers of 0.5-mm polyvinyl chloride (PVC) and one layer of 1.5-mm thick fiber to increase strength of foot orthoses in the bottom layers as well as one layer of 1.2-mm genuine leather in the upper layer to increase comfort.
  The participants will be asked to use the CFO in daily life during weight-bearing activities.
  Arms: Insole group

SUMMARY:
Plantar heel pain (PHP), normally known as plantar fasciitis, is a common encountered musculoskeletal problem in the foot that can cause activities limitation, difficulty, and discomfort especially while standing and walking. It involves pain and inflammation of the plantar fascia, which runs across the bottom of the foot and connects the heel bone to toes. Approximately 10% of the American population have inferior heel pain in their lifetime, and 80% in these patients were diagnosed as the PHP.

According to Sullivan's study, they identified the musculoskeletal factors in PHP and found that the ankle evertors, peroneus brevis and longus muscles, and toe flexors, flexor hallucis longus and brevis muscles, flexor digitorum longus and brevis muscles were weaker than the normal. Moreover, previous studies reported that the patients with PHP frequently have weakness of the tibialis posterior muscle.

Since the presence of PHP involved with the deviation of lower-extremity biomechanics, foot orthoses have been the common intervention used as a part of the conservative treatment. The previous cadaveric study provided helpful information regarding the mechanism of foot orthoses; the researchers explained that foot orthoses could reduce plantar fascia strain during stance phase by lifting the medial longitudinal arch and decreasing abnormal foot pronation. Therefore, custom-fitted orthoses should be used to provide individual comfort, maintain the height of medial longitudinal arch, and also protect the excessive tensile strain of the plantar fascia.

Therefore, the present study interested to compare the effectiveness of home based strengthening exercise program and the low-cost CFO on pain intensity, foot function, and lower-extremity biomechanics during walking in patients with PHP.

DETAILED DESCRIPTION:
PHP can be presented with a high prevalence in both athletic and non-athletic populations. Diagnosis of the PHP based on patients' history and physical examination. To obtain the correct diagnosis of the PHP, subjective and objective physical examinations should be performed.

PHP is believed that it occurs from the excessive cumulative strain of the plantar fascia enthesis or the insertion of the plantar fascia. This excessive strain resulted in repetitive microtrauma or inflammatory condition. Sullivan in 2015, studied musculoskeletal and activity factors that associated with PHP. The results showed that the impairments in patients with PHP have a high association with high body mass index (BMI), decrease in ankle dorsiflexion range of motion (ROM), and weakness of ankle evertors and toe flexors muscles. Therefore, these factors may have a high chance to induce the recurrence of PHP.

The PHP management could be approached either surgical or non-surgical treatment. The previous studies showed conflict and fewer evidences ineffectiveness of the treatment for PHP. Moreover, approximately 18 - 50% of patients with PHP who received conservative treatment still presenting their symptoms and pain in 2 years after diagnosis and 30% have recurrent PHP. From the above-mentioned review, there are few studies investigating the effect of strengthening exercise for the foot and ankle muscles on PHP.

The weakness of foot and ankle muscles may lead to recurrent symptoms of PHP due to insufficient muscle function, co-contraction of muscles, and foot joints position during walking. Thus, peroneus brevis and longus muscles, tibialis posterior muscles, flexor hallucis longus and brevis muscles, flexor digitorum longus and brevis muscles should be strengthening.

As described in American clinical practice guideline, customized foot orthoses (CFO) could be used to provide short-term management (3 months) for pain reduction and foot function improvement. Among all conservative options, CFO is routinely used in clinical practice and widely recommended.

ELIGIBILITY:
Inclusion Criteria:

* Reaching the specific criteria of PHP including (15)

  * A complaint of tenderness from the palpation of the medial calcaneal tubercle and the medial aspect of the proximal portion of the plantar fascia, or pain along the plantar fascia at medial longitudinal arch side
  * The presence of heel pain immediately during the first few steps of walking in the morning or after prolonged period of inactivity; and gradually decreased throughout the day with ordinary walking; and worsened with prolonged activity
* Having the symptom of heel pain for at least 6 weeks, indicating the chronic condition (29)
* Having maximum level of pain intensity during last week using visual analog scale (VAS) ranging from 3 to 6 mm

Exclusion Criteria:

* Having BMI more than 30 kg/m2 (40)
* Having leg length difference more than 1 cm (30)
* Unable to perform the exercise program
* Having positive sciatica test, indicating the L5-S1 nerve root irritation
* Having history of lower extremity fracture
* Having history of lower extremity surgery
* Having been diagnosed with gout, diabetic neuropathy, rheumatoid arthritis, systemic lupus erythematosus (SLE), cancer, infection disease and tumor

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 70 (Estimated)
Dates: Start 2021-04-01 (Actual); Primary Completion 2023-09-30 (Estimated); Study Completion 2023-09-30 (Estimated)

PRIMARY OUTCOMES:
Pain at Worst | End of 3rd month
  The participants were asked about pain at the worst in the past week. Visual analogue scale (VAS) was used for the participants to rate the pain on the paper with the 10 centimeters (cm) line. Left and right ends of the line demonstrate "no pain with 0 score" and "worst pain ever with 10 scores".

SECONDARY OUTCOMES:
Foot Function Score | baseline, end of 1st month, end of 2nd month, and end of 3rd month
  The Foot Function Index (FFI) is a self-rating questionnaire that reflexes the foot health via pain and function (45-47). It consists of the 23 questions of the difficulty level and pain during performing foot function with the visual analogue scale for each question. The score ranges from 0-230 and minimum score represents a good condition of foot pain and function. This study used the Thai version of FFI that translated forward and backward from the English version.
Plantar Fascia Thickness | baseline, end of 1st month, end of 2nd month, and end of 3rd month
  Plantar fascia thickness was assessed by using a portable digital Ultrasound (US) diagnosis imaging system, D-6600 (Mindray, China) with a 10 MHz wideband linear array probe, operate by the researcher. Test-retest reliability was proved and showed excellent reliability at ICC 0.969 (Appendix I). To evaluate the plantar fascia thickness, scan depth was set at 4 cm (48, 49). The researcher assessed the thickness on the symptomatic foot of the participants or the most painful side in patients with bilateral PHP.
Gait assessment | baseline, end of 1st month, end of 2nd month, and end of 3rd month
  Gait assessment will be performed at the motion analysis research laboratory of the Faculty of Physical Therapy, Mahidol University. This laboratory consists of an eight-camera motion analysis system (Motion Analysis Corporation, Santa Rosa, CA, USA) with a sample rate of 120 Hz. The cameras are synchronized with three force transducers (Bertec force plate, Columbus, OH, USA), which are set to have a sample rate of 1200 Hz on a 10-meter walkway. The software for the motion analysis system is CORTEX version 2.5 with three major functions consisting of calibration of capture volume, tracking and identifying marker locations in calibrated 3D space, and post-processing tools for tracking, editing, and preparing data for other packages. Marker histories and analog signals are smoothed with a 6th order, low-pass Butterworth filter at 5 Hz and 50 Hz, respectively.
Pain at Worst | baseline, end of 1st month, and end of 2nd month
  The participants were asked about pain at the worst in the past week. Visual analogue scale (VAS) was used for the participants to rate the pain on the paper with the 10 centimeters (cm) line. Left and right ends of the line demonstrate "no pain with 0 score" and "worst pain ever with 10 scores".

CONTACTS AND LOCATIONS:
Overall Officials: Suthasinee Thong-On, PhD, Principal Investigator — Dr.
Locations (1):
- Faculty of Physical Therapy, Mahidol University, Nakhon Pathom, Thailand

IPD SHARING:
Plan to Share IPD: No
No sharing of the data.